CLINICAL TRIAL: NCT05772234
Title: Aggressive Intravenous Hydration With Lactated Ringer's Solution for Prevention of Post-ESWL Pancreatitis: A Multicenter, Prospective, Randomized Clinical Trial
Brief Title: Aggressive Intravenous Hydration With Lactated Ringer's Solution for Prevention of Post-ESWL Pancreatitis
Acronym: HYPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Ruijin Hospital (Other); LanZhou University (Other); First People's Hospital of Hangzhou (Other); The Second Affiliated Hospital of Baotou Medical College (Other); Shanghai Pudong New Area Gongli Hospital (Other); Peking Union Medical College Hospital (Other); Qilu Hospital of Shandong University (Other); The Third Xiangya Hospital of Central South University (Other); Affiliated Hospital of Yunnan University (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HYPER20221204
Record Dates: First submitted 2023-02-18; First posted 2023-03-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Pancreatitis, Chronic; Pancreatic Duct Stone
Keywords: pancreatic extracorporeal shock wave lithotripsy; post-ESWL pancreatits; intravenous hydration; lactated Ringer's solution
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aggressive hydration group (Experimental): Periprocedural hydration with intravenous 20 mL/kg lactated Ringer's solution within 60 min from the start of ESWL (first shockwave delivered), directly followed by 3 mL/kg per h for 8 h.
  Interventions: Drug: Lactated ringers solution
- Restricted hydration group (Active Comparator): Periprocedural hydration with normal saline (maximum of 1.5mL/kg per h or 3L per 24h).
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Lactated ringers solution — Intravenous 20 mL/kg Ringer's lactate solution within 60 min from the start of ESWL, directly followed by 3 mL/kg per h for 8 h.
  Arms: Aggressive hydration group
Drug: normal saline — Intravenous fluid infusion with normal saline (maximum of 1.5mL/kg per h or 3L per 24h).
  Arms: Restricted hydration group

SUMMARY:
The goal of this clinical trial is to clarify whether aggressive intravenous hydration with lactated Ringer's solution could reduce the incidence of post-ESWL pancreatitis in patients with chronic pancreatitis.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is a disease caused by genetic and environmental factors that lead to progressive fibrosis of the pancreatic tissue, resulting in irreversible damage to the structure and function of the pancreas. The incidence of pancreatic duct stones in CP is as high as 90%. Stones can lead to pancreatic duct obstruction, pancreatic parenchymal hypertension and ischemia, inducing frequent abdominal pain and accelerating the decline of pancreatic function, therefore, removal of pancreatic duct stones is important for relieving CP symptoms. For large stones and complex stones, pancreatic extracorporeal shock wave lithotripsy (P-ESWL) was recommended. Acute pancreatitis is the most common complication after P-ESWL with an incidence of 6.3-12.5%, which result in prolonged hospitalization, increased medical costs, and can be life-threatening.

There are few studies on the prevention of postoperative pancreatitis after P- ESWL. Only one prospective randomized controlled study found the role of NSAIDs in the prevention of acute pancreatitis after ESWL, and preoperative use of rectal indomethacin reduced post-ESWL pancreatitis from 12% to 9%. ERCP placement of pancreatic duct stent is one of the effective methods to prevent post-ERCP pancreatitis. However, studies have shown that pancreatic duct stenting before ESWL is not effective in preventing acute pancreatitis after P-ESWL. More research is needed in the prevention and treatment of pancreatitis after P-ESWL.

There have been more high-quality studies on the prevention of post-ERCP pancreatitis. In addition to NSAIDs, several prospective randomized controls have found that perioperative high-dose lactated Ringerolysis (LRS) hydration is effective in preventing acute pancreatitis after ERCP. In a meta-analysis, active hydration of LRS was found to reduce post-ERCP pancreatitis from 13% to 6%. Based on above findings, international guidelines recommend aggressive perioperative LRS hydration to reduce the risk of post-ERCP pancreatitis.

Previous studies have suggested various mechanisms leading to post-ERCP pancreatitis, including mechanical injury, chemical injury, hydrostatic injury, and infection. Given the potentially similar pathogenesis of postoperative pancreatitis, we propose to conduct a randomized controlled trial to investigate the efficacy of active hydration of lactated Ringer's solution for the prevention of post-ESWL pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

All patients with chronic pancreatitis aged between18 and 85 years who were eligible for treatment with ESWL for pancreatic stones were eligible for enrolment.

Exclusion Criteria:

1. Patients readmitted to the hospital for ESWL during the study period.
2. Acute pancreatitis in the last 3 days.
3. Signs of congestive heart failure, such as pitting edema or a New York Heart Association classification greater than class I heart failure. For patients ≥ 70 years old, brain natriuretic peptide (BNP) and cardiac ultrasound would be performed before ESWL. Patients with BNP>100pg/ml or Ejection Fraction value<50% should be excluded.
4. Respiratory insufficiency (pO2 < 60 mmHg or saturation < 90% despite FiO2 of 30% or requiring mechanical ventilation). For patients ≥ 70 years old, pulmonary function tests would be performed before ESWL. Patients with Forced Expiratory Volume in the first second (FEV1) <70% are excluded.
5. Severe liver disease (cirrhosis, liver abscess).
6. Patients receiving more than 1.5 mL/kg/h or 3 L/24 h of intravenous fluids in the 24 h before ESWL.
7. Hypotension (systolic blood pressure <90 mmHg or mean arterial pressure <70 mmHg).
8. Hypo- or hypernatremia (serum Na+ levels < 130 or > 150 mmol/L).
9. Pregnancy.
10. Unwilling or unable to provide consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1066 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of post-ESWL pancreatitis | 24 hours
  Post-ESWL pancreatitis is defined according to the 2012 Atlanta criteria. A diagnosis of post-ESWL pancreatitis is made if two of three of the following criteria are met: pain consistent with pancreatitis; amylase or lipase of at least three times the upper normal limit within 24 h of the procedure; or characteristic findings on imaging.

SECONDARY OUTCOMES:
Severity of pancreatitis | 1 month
  Stratified as mild, moderate, or severe, mainly on the basis of length of hospitalization and need for invasive treatment.
Incidence of other post-ESWL complications | 24 hours
  Including bleeding, infection, steinstrasse, and perforation.
Incidence of fluid overload | 24 hours
  Including pulmonary or peripheral edema and congestive heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Lianghao Hu, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] Buxbaum JL, Freeman M, Amateau SK, Chalhoub JM, Coelho-Prabhu N, Desai M, Elhanafi SE, Forbes N, Fujii-Lau LL, Kohli DR, Kwon RS, Machicado JD, Marya NB, Pawa S, Ruan WH, Sheth SG, Thiruvengadam NR, Thosani NC, Qumseya BJ; (ASGE Standards of Practice Committee Chair). American Society for Gastrointestinal Endoscopy guideline on post-ERCP pancreatitis prevention strategies: summary and recommendations. Gastrointest Endosc. 2023 Feb;97(2):153-162. doi: 10.1016/j.gie.2022.10.005. Epub 2022 Dec 12. No abstract available. PMID 36517310
- [Background] Skolarikos A, Alivizatos G, de la Rosette J. Extracorporeal shock wave lithotripsy 25 years later: complications and their prevention. Eur Urol. 2006 Nov;50(5):981-90; discussion 990. doi: 10.1016/j.eururo.2006.01.045. Epub 2006 Feb 7. PMID 16481097
- [Background] Li BR, Liao Z, Du TT, Ye B, Zou WB, Chen H, Ji JT, Zheng ZH, Hao JF, Jiang YY, Hu LH, Li ZS. Risk factors for complications of pancreatic extracorporeal shock wave lithotripsy. Endoscopy. 2014 Dec;46(12):1092-100. doi: 10.1055/s-0034-1377753. Epub 2014 Sep 24. PMID 25251205
- [Background] Tandan M, Nageshwar Reddy D, Talukdar R, Vinod K, Kiran SVVS, Santosh D, Gupta R, Ramchandani M, Lakhtakia S, Rakesh K, Manohar Reddy P, Basha J, Nabi Z, Jagtap N, Rao GV. ESWL for large pancreatic calculi: Report of over 5000 patients. Pancreatology. 2019 Oct;19(7):916-921. doi: 10.1016/j.pan.2019.08.001. Epub 2019 Aug 2. PMID 31447280
- [Background] Qian YY, Ru N, Chen H, Zou WB, Wu H, Pan J, Li B, Xin L, Guo JY, Tang XY, Hu LH, Jin ZD, Wang D, Du YQ, Wang LW, Li ZS, Liao Z. Rectal indometacin to prevent pancreatitis after extracorporeal shock wave lithotripsy (RIPEP): a single-centre, double-blind, randomised, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2022 Mar;7(3):238-244. doi: 10.1016/S2468-1253(21)00434-9. Epub 2022 Jan 25. PMID 35085482
- [Background] Choi JH, Kim HJ, Lee BU, Kim TH, Song IH. Vigorous Periprocedural Hydration With Lactated Ringer's Solution Reduces the Risk of Pancreatitis After Retrograde Cholangiopancreatography in Hospitalized Patients. Clin Gastroenterol Hepatol. 2017 Jan;15(1):86-92.e1. doi: 10.1016/j.cgh.2016.06.007. Epub 2016 Jun 14. PMID 27311618
- [Background] Park CH, Paik WH, Park ET, Shim CS, Lee TY, Kang C, Noh MH, Yi SY, Lee JK, Hyun JJ, Lee JK. Aggressive intravenous hydration with lactated Ringer's solution for prevention of post-ERCP pancreatitis: a prospective randomized multicenter clinical trial. Endoscopy. 2018 Apr;50(4):378-385. doi: 10.1055/s-0043-122386. Epub 2017 Dec 13. PMID 29237204
- [Background] Sperna Weiland CJ, Smeets XJNM, Kievit W, Verdonk RC, Poen AC, Bhalla A, Venneman NG, Witteman BJM, da Costa DW, van Eijck BC, Schwartz MP, Romkens TEH, Vrolijk JM, Hadithi M, Voorburg AMCJ, Baak LC, Thijs WJ, van Wanrooij RL, Tan ACITL, Seerden TCJ, Keulemans YCA, de Wijkerslooth TR, van de Vrie W, van der Schaar P, van Dijk SM, Hallensleben NDL, Sperna Weiland RL, Timmerhuis HC, Umans DS, van Hooft JE, van Goor H, van Santvoort HC, Besselink MG, Bruno MJ, Fockens P, Drenth JPH, van Geenen EJM; Dutch Pancreatitis Study Group. Aggressive fluid hydration plus non-steroidal anti-inflammatory drugs versus non-steroidal anti-inflammatory drugs alone for post-endoscopic retrograde cholangiopancreatography pancreatitis (FLUYT): a multicentre, open-label, randomised, controlled trial. Lancet Gastroenterol Hepatol. 2021 May;6(5):350-358. doi: 10.1016/S2468-1253(21)00057-1. Epub 2021 Mar 19. PMID 33740415
- [Background] Wu BU, Hwang JQ, Gardner TH, Repas K, Delee R, Yu S, Smith B, Banks PA, Conwell DL. Lactated Ringer's solution reduces systemic inflammation compared with saline in patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):710-717.e1. doi: 10.1016/j.cgh.2011.04.026. Epub 2011 May 12. PMID 21645639
- [Background] Radadiya D, Devani K, Arora S, Charilaou P, Brahmbhatt B, Young M, Reddy C. Peri-Procedural Aggressive Hydration for Post Endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis Prophylaxsis: Meta-analysis of Randomized Controlled Trials. Pancreatology. 2019 Sep;19(6):819-827. doi: 10.1016/j.pan.2019.07.046. Epub 2019 Jul 30. PMID 31383573